CLINICAL TRIAL: NCT01220206
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Design Trial to Evaluate the Safety and Efficacy of POM Wonderful Pomegranate Extract Capsules In Male Subjects With Moderate to Severe Erectile Dysfunction
Brief Title: POMx In the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: POM Wonderful LLC (Industry)
Collaborators: Target Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POM 2010-003
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Erectile Dysfunction
Keywords: ED; POMx; Pomegranate; Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 2 placebo capsules daily
  Interventions: Drug: Placebo
- one POMx capsule (Experimental): One POMx capsule, one placebo capsule daily
  Interventions: Drug: One POMx capsule daily
- 2 POMx Capsules (Experimental): 2 POMx Capsules daily
  Interventions: Drug: 2 POMx Capsules

INTERVENTIONS:
Drug: Placebo — 2 placebo capsules daily
  Arms: Placebo
Drug: One POMx capsule daily — One POMx capsule, one placebo capsule daily
  Arms: one POMx capsule
Drug: 2 POMx Capsules — 2 POMx Capsules daily
  Arms: 2 POMx Capsules

SUMMARY:
POMx can be used as a treatment for erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male 21 to 70 years old
* Erectile Function domain score of 10-19 on the International Index of Erectile Function (IIEF)
* In a stable, monogamous relationship with a consenting female partner and willing to attempt vaginal sexual intercourse on at least one occasion per week on average during each study period
* History of ED (clinically defined as the inability to attain and maintain an erection of the penis sufficient to permit satisfactory sexual intercourse) of at least 3 months duration
* Treated previously with a PDE-5 inhibitor with a satisfactory response, as defined by the patient.
* Signed informed consent

Exclusion Criteria:

-The presence of any of the following excludes a subject from study enrollment: ED caused by untreated endocrine disease, i.e., hypopituitarism, hypothyroidism, hypogonadism

* A diagnosis of situational psychogenic ED
* Significant penile pathology, including but not limited to curvature, fibrosis, sexually transmitted disease, and penile implant
* Clinically significant hepatic, renal, neurological disease, diabetes mellitus, spinal cord injury, significant coronary heart disease, significant neurological disease or hepatitis B and/or C
* History of prostate cancer or prostate surgery other than a transurethral resection of the prostate
* History of alcoholism within the previous 2 years
* Current consumer of three or more units of alcohol per day (1 unit is equivalent to 1 glass of wine, 1 pint of beer, or 1 shot of hard liquor)
* Taking ED therapy (prescription medications, over-the-counter medications, herbal preparations or medical devices) after the screening visit
* Participation in another study with an investigational drug or device during the 30 days prior to study entry
* Has a condition interfering with his ability to provide informed consent or comply with study instructions

Ages: 21 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Effects on ED | Basedline to end of study
  There are three co-primary endpoints: Erectile Function domain score (questions 1-5 and 15 of the IIEF), and questions 2 and 3 on the SEP diary

SECONDARY OUTCOMES:
Effect on ED | baseline to end of study
  Secondary efficacy variables are: Total score on SEP and domains of the IIEF representing intercourse satisfaction (questions 6-8), orgasmic function (questions 9-10), and overall satisfaction (questions 11-12) and a Global Assessment Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: James McMurray, MD, Principal Investigator — Medical Affiliated Research Center, Inc.
Locations (1):
- Medical Affiliated Research Center, Huntsville, Alabama, United States